CLINICAL TRIAL: NCT02307422
Title: Genetic Polymorphisms Associating With CAD, Inflammatory Biomarkers, and Oxidized Phospholipids in a Greek Population
Brief Title: Genetic Polymorphisms Associated With CAD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Interleukin Genetics, Inc. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Other Study IDs: ILI-14-133-C-UCSD
Record Dates: First submitted 2014-11-21; First posted 2014-12-04 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — DNA has been extracted from previously obtained subject blood samples at the University General Hospital of Ioannina, Greece study site. DNAs will be labeled by anonymized subject ID # (de-identified), and shipped to ILI for genotyping and genetic analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Diabetic patients undergoing coronary angiography (both sexes), who are age 18-90, and admitted in the Department of Cardiology in the University General Hospital of Ioannina and Catheterization Laboratory of 1st IKA Hospital in Athens and undergo coronary angiography for clinical purposes will be studied. Presence epicardial vessel stenosis (>50%), and multi-vessel disease will be recorded. Excluded: previous history of revascularization procedure or moderate to severe stenosis. Patient samples will be evaluated for quantitative levels of the biomarkers Lp(a) and OXPL/apoB. IL-1 Genotypes, and other SNPs associated with CAD will be assessed in this group and related to levels of Lp(a) and oxidized phospolipids. No interventions other than the post-hoc DNA testing will be performed.
  Interventions: Genetic: IL-1 Genotypes, other SNPs associated with CAD
- Control: Non-diabeticpatients undergoing coronary angiography (both sexes), who are age 18-90, and admitted in the Department of Cardiology in the University General Hospital of Ioannina and Catheterization Laboratory of 1st IKA Hospital in Athens and undergo coronary angiography for clinical purposes will be studied. Presence epicardial vessel stenosis (>50%), and multi-vessel disease will be recorded. Excluded: previous history of revascularization procedure or moderate to severe stenosis. Patient samples will be evaluated for quantitative levels of the biomarkers Lp(a) and OXPL/apoB. IL-1 Genotypes, and other SNPs associated with CAD will be assessed in this group and related to levels of Lp(a) and oxidized phospolipids. No interventions other than the post-hoc DNA testing will be performed.
  Interventions: Genetic: IL-1 Genotypes, other SNPs associated with CAD

INTERVENTIONS:
Genetic: IL-1 Genotypes, other SNPs associated with CAD — Genotyping will be carried out by a CLIA-certified genotyping facility at ILI, Waltham MA. DNA concentrations will be adjusted to a range compatible with multiple PCR conditions. Genotyping will be accomplished by performing multiplex polymerase chain reactions (PCR) specifically targeting the surrounding sequences for the SNPs being studied. A single base extension assay will be hybridized to a 48-plex microarray plate and read on a SNPstream Genotyping System (Beckman-Coulter).

SUMMARY:
The design and purpose of the current study is to expand and validate previous findings that the IL-1 gene cluster composite genotype patterns potentiate the risk for coronary artery disease (CAD) and cardiovascular events mediated by OxPL and Lp(a). A secondary objective is to validate other, non IL-1 genetic variants associated with CAD.

DETAILED DESCRIPTION:
The conclusions from an earlier study indicate that the contribution of OxPL/apoB and Lp(a) on angiographically documented CAD and CAD events is conditional on proinflammatory IL-1 genotypes. This novel paradigm links the etiology of atherogenesis attributed to OxPL and Lp(a) from genetics to clinical expression of CAD. ILI has also identified the functional IL-1 gene variations that regulate the IL1B gene in a haplotype context and appear to explain over-expression of IL-1β, as well as the expression of other inflammatory biomolecules that are downstream of IL-1β. The functional IL-1 variants have been combined into patterns that have been associated with risk for more severe periodontal disease across multiple ethnic/racial populations. It is also important to test this functional genetic pattern for similar interactions with OxPL and Lp(a) biomarker levels in association with angiographically documented CAD and CAD events. DNA has been extracted from previously obtained subject blood samples (1173 subjects; 18 years to 90 years at entry (coronary angiography)) at the University General Hospital of Ioannina, Greece study site. DNAs will be labeled by anonymized subject ID # (de-identified), and shipped to ILI for genotyping and genetic analysis. Phase II will determine whether other gene variations (SNPs) previously shown in the literature to be associated with CAD and/or CAD-related secondary events can be validated in this study population.

ELIGIBILITY:
Inclusion Criteria: Diabetics and non-diabetics, with or without known CV disease, who are admitted in the Department of Cardiology in the University General Hospital of Ioannina and the Catheterization Laboratory of 1st IKA Hospital in Athens and undergo coronary angiography at ages 18-90 for clinical purposes will be studied. The study includes subjects who; 1) have suspected CAD and undergo a scheduled diagnostic angiogram for clinical reasons, and 2) are hospitalized because of an acute coronary syndrome and thus undergo diagnostic angiography (with or without previous history of CAD).

-

Exclusion Criteria: Patients < 18 years old and > 90 years old at time of coronary angiography. Patients with a previous history of coronary revascularization procedure or moderate to severe stenosis will be excluded.

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between 18 years to 90 years at entry (coronary angiography) of both genders. Patients with a previous history of coronary revascularization procedure or moderate to severe stenosis will be excluded. Diabetics and non-diabetics, with or without known CV disease, who are admitted in the Department of Cardiology in the University General Hospital of Ioannina and the Catheterization Laboratory of 1st IKA Hospital in Athens and undergo coronary angiography for clinical purposes will be studied. The study includes subjects who; 1) have suspected CAD and undergo a scheduled diagnostic angiogram for clinical reasons, and 2) are hospitalized because of an acute coronary syndrome and thus undergo diagnostic angiography (with or without previous history of CAD).
Sampling Method: Probability Sample
Enrollment: 1173 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Evidence of IL-1 risk genotypes of the Heart Health Test in relation to levels of Lp(a)(mg/dL) and oxPL/apoB (RLU) in CAD patients. | Approximately 1 year
  Compare the frequencies of positive and negative genetic test results (Heart Health Test, composite genotype of rs17561, rs1143634, rs16944) among CAD patients based on previously collected levels (eg. quartiles) of LP(a) and specific oxidized phospholipids among diabetic and non-diabetic subjects.

SECONDARY OUTCOMES:
Evidence of IL-1 risk genotypes of the PerioPredict Test in relation to levels of Lp(a)(mg/dL) and oxPL/apoB (RLU) in CAD patients. | Approximately 1 year
  Compare the frequencies of positive and negative genetic test results (PerioPredict Test, composite genotype of rs16944, rs1143623, rs4848306, rs1143633)among CAD patients based on previously collected levels (eg. quartiles) of LP(a) and specific oxidized phospholipids among diabetic and non-diabetic subjects.
Evidence for other non IL-1 gene SNPs, previously shown to be associated with CAD, in relation to levels of Lp(a)(mg/dL) and oxPL/apoB (RLU) among diabetic and non-diabetic patients. | Approximately 1 year
  Compare the frequencies of SNP alleles, haplotypes, and composite genotypes among CAD patients based on levels (eg. quartiles) of LP(a) in mg/dL and oxidized phospholipids/apoB (RLU) among diabetic to non-diabetic subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Doucette-Stamm, Ph.D., Study Director — Interleukin Genetics, Inc.

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with collaborators at University of California San Diego, La Jolla, California.

REFERENCES:
- [Background] Tsimikas S, Duff GW, Berger PB, Rogus J, Huttner K, Clopton P, Brilakis E, Kornman KS, Witztum JL. Pro-inflammatory interleukin-1 genotypes potentiate the risk of coronary artery disease and cardiovascular events mediated by oxidized phospholipids and lipoprotein(a). J Am Coll Cardiol. 2014 May 6;63(17):1724-34. doi: 10.1016/j.jacc.2013.12.030. Epub 2014 Feb 12. PMID 24530664